CLINICAL TRIAL: NCT06996587
Title: A Randomized Controlled Trial Comparing Efficacy, Ergonomics, and Safety of ILY Robotic System vs Manual Flexible Ureteroscopy in Patients Undergoing Laser Lithotripsy for Kidney Stones
Brief Title: ILY Robotic System vs Manual Flexible Ureteroscopy for Kidney Stone Treatment
Acronym: iFURS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert El Hajj (Other)
Responsible Party: Sponsor-Investigator, Albert El Hajj, Associate Professor of Urology, American University of Beirut Medical Center
Organization: American University of Beirut Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2024-0452
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stones; Urolithiasis
Keywords: kidney stones; manual flexible ureteroscopy; fURS; ILY robot; robotic
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic-Assisted fURS Group using the ILY Robot (Experimental): Participants undergo flexible ureteroscopy using the ILY® robotic system.
  Interventions: Procedure: Robotic-Assisted Flexible Ureteroscopy
- Manual fURS Group (Active Comparator): Participants undergo standard manual flexible ureteroscopy.
  Interventions: Procedure: Manual Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Robotic-Assisted Flexible Ureteroscopy — Use of the ILY® robotic system to perform flexible ureteroscopy.
  Arms: Robotic-Assisted fURS Group using the ILY Robot
Procedure: Manual Flexible Ureteroscopy — Conventional flexible ureteroscopy performed manually by the surgeon.
  Arms: Manual fURS Group

SUMMARY:
The goal of this clinical trial is to compare the efficacy, ergonomics, and safety of robotic versus manual flexible ureteroscopy (fURS) for kidney stone treatment in adult patients undergoing laser lithotripsy.

* Does robotic-assisted lithotripsy using the ILY® robot have the same efficacy as the manual fURS in treating kidney stones?
* Is robotic flexible ureteroscopy associated with similar or improved safety outcomes, including perioperative and 30-day postoperative complication rates?
* Does the robotic system offer improved ergonomics, lower surgeon radiation exposure, and favorable intraoperative metrics compared to manual flexible ureteroscopy? Researchers will compare the ILY robotic system with manual fURS to see if robotic intervention can match or improve clinical and ergonomic outcomes.

Participants will:

* Be randomly assigned to undergo laser lithotripsy with either the ILY robot or manual flexible ureteroscopy
* Complete standard pre- and postoperative assessments
* Undergo evaluation for stone-free status using a non-contrast CT scan at 30 days postoperatively
* Undergo evaluation for postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 years old
* Patients with a normal pelvicalyceal anatomy
* Patients with renal stone diagnosis confirmed by noncontrast computed tomography regardless of stone size, location, and multiplicity
* ASA score I-III
* Intact mental and cognitive ability to provide informed consent and willingness to participate in the study with 30-day follow-up

Exclusion Criteria:

* Children < 18 and pregnant women
* Patients with anatomically anomalous kidneys, known case of stricture or stenosis, or recent 3-month history of ureteroscopy (DJ stent placement only will be accepted) or known history of complicated ureteroscopy
* Patients in whom stone measurement was not feasible on NCCT or those with concomitant ureteric stones.
* ASA score IV
* Mentally incapacitated patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy assessed by measuring the stone-free rate (SFR) | 30 days after the index procedure
  A patient is considered stone free if there are no visible residual stone fragments after the treatment.

SECONDARY OUTCOMES:
Perioperative and 30-day Postoperative Outcomes | Perioperatively and 30 days after the procedure
  This assessment will account for any complications related to the patient's clinical condition from the procedure through a 4-week postoperative period.
Ergonomics | Immediately after the procedure
  The NASA Task Load Index will be used to assess for ergonomics.
Surgeon safety in terms of radiation exposure | During the procedure
  Surgeon safety from ionizing radiation will be assessed by the surgeon wearing 3 dosimeter badges used to detect and record exposure.
Intraoperative Parameters | During the procedure
  Operative time, draping time, docking time, lasing time (all measured in minutes)
Conversion rate | During the procedure
  The proportion of cases where a procedure originally planned using the robotic technique had to be converted to manual fURS due to complications, technical difficulties, or failure of equipment.

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Coded participant data, including baseline characteristics, primary and secondary outcome measures, and statistical analysis plans will be made available upon reasonable request from the corresponding author. The study protocol, statistical analysis plan, and informed consent forms will also be accessible upon request. Researchers seeking data must submit a methodologically sound proposal, which will be reviewed by the trial steering committee. Data will be shared in compliance with institutional and ethical regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning six months after publication and ending five years after the publication date

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT06996587/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT06996587/ICF_001.pdf